CLINICAL TRIAL: NCT02814396
Title: The Application of Multichannel ECG Analytic System in Cardiovascular Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201207070RIC
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2023-04

CONDITIONS: Multichannel ECG System
Keywords: Ventricular; CVD; Ventricular arrhythmias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death worldwide. Most individuals with CVD show no evidence of disease for decades as the disease progresses before the first onset of symptoms, often a "sudden" heart attack, finally arises. The spatial repolarization heterogeneity within the ventricular myocardium had been proposed to represent the function of the heart in health and disease. Greater than normal levels of repolarization dispersion may allow early diagnosis of CVD. There is a growing interest in the characteristic features of ventricular repolarization that leads to lethal ventricular arrhythmia even with the use of non-antiarrhythmic drugs. The recovery time dispersion may reflect a repolarization heterogeneity leading to lethal ventricular arrhythmia. Previously, the investigators had utilized a 64-channel low-TC SQUID MCG device to develop and verify 2 parameters, so called smooth index of QTc (SIQTc) and T wave propagation (TWP), to accurately detect and localize the myocardial ischemia. Recently Nakai, et al. reported that a newly developed 187-ch signal-averaged vector-projected ECG (187-ch SAVP-ECG) could evaluate low-amplitude high-frequency potentials and repolarization heterogeneity. In this project, the investigators'll try to modify and improve the spatial resolution of ECG signals from a Self-built-in multichannel ECG system with a newly developed algorithm, and also try to derive the SIQTc and TWP from this system, for early detection of CVD. The investigators intend to prove the concept that this newly developed multichannel ECG system could efficiently detect or diagnose CVD with acceptable sensitivity and specificity, and in a portable way.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death worldwide. Most individuals with CVD show no evidence of disease for decades as the disease progresses before the first onset of symptoms, often a "sudden" heart attack, finally arises. The spatial repolarization heterogeneity within the ventricular myocardium had been proposed to represent the function of the heart in health and disease. Greater than normal levels of repolarization dispersion may allow early diagnosis of CVD. There is a growing interest in the characteristic features of ventricular repolarization that leads to lethal ventricular arrhythmia even with the use of non-antiarrhythmic drugs. The recovery time dispersion may reflect a repolarization heterogeneity leading to lethal ventricular arrhythmia. Although cheap and convenient, the traditional 12-leads electrocardiogram (ECG) is frequently normal at rest in such patients. The quantification of repolarization heterogeneity with ECG, QT dispersion, has some methodological limitations and has been abandoned in daily practice. Many studies have shown that body surface potential mapping (BSPM) contains more diagnostic and prognostic information than that elicited from a 12-lead ECG. The BSPM and magnetocardiogram (MCG) are two new developed recording methods, and provide higher spatial resolution than traditional ECG signals but with the disadvantages of high cost and huge volume. It is impossible to be used in a portable way. Previously, the investigators had utilized a 64-channel low-TC SQUID MCG device to develop and verify 2 parameters, so called smooth index of QTc (SIQTc) and T wave propagation (TWP), to accurately detect and localize the myocardial ischemia. Recently Nakai, et al. reported that a newly developed 187-ch signal-averaged vector-projected ECG (187-ch SAVP-ECG) could evaluate low-amplitude high-frequency potentials and repolarization heterogeneity. In this project, the investigators'll try to modify and improve the spatial resolution of ECG signals from a Self-built-in multichannel ECG system with a newly developed algorithm, and also try to derive the SIQTc and TWP from this system, for early detection of CVD. The investigators intend to prove the concept that this newly developed multichannel ECG system could efficiently detect or diagnose CVD with acceptable sensitivity and specificity, and in a portable way.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years old.
* with suspected arrhythmia or cardiovascular diseases.

Exclusion criteria

* NO

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Space ventricular repolarization within the proposal does not have to represent functions in heart health and disease. Repolarization dispersion higher than normal levels may allow early diagnosis of CVD.
  The BSPM and magnetic diagram (MCG) is a newly developed method for both records, and provide higher spatial resolution than conventional ECG signal but has a high cost and bulky shortcomings. It is impossible in a portable manner. Previously, the investigators have used a 64-channel low TC SQUID MCG equipment to develop and validate two parameters, the so-called QT interval (SIQTc) and T wave propagation (TWP) smoothness index, accurate detection and localization of myocardial ischemia blood.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-01; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Composite cardiovascular outcome | up to 5 years
  The composite cardiovascular (CV) outcome will be any CV events (coronary, cerebral, or peripheral vascular diseases)

SECONDARY OUTCOMES:
With at least 1 cardiovascular risk factor. | up to 5 years
  no evidence of atherosclerotic vascular diseases,with at least 1 cardiovascular risk factor.

CONTACTS AND LOCATIONS:
Overall Officials: Chau C WU, M.D.,Ph.D., Principal Investigator — chauchungwu@ntu.edu.tw
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes